CLINICAL TRIAL: NCT02210585
Title: Study of Multi-site Neuromuscular Electrical Stimulation to Increase Spontaneous Physical Activity in Obesity Patient Carrying Severe Inactive: Randomized Controlled Trial vs Placebo
Brief Title: Study of Neuromuscular Electrical Stimulation to Increase Spontaneous Physical Activity in Obesity Patient
Acronym: STIMOBIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38RC13.554
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Number of Steps Per Day < 7000
MeSH Terms: conditions — Obesity | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kneehab® (Active Comparator): 5 sessions per week
  Interventions: Other: Rehabilitation
- Placebo (Placebo Comparator): 5 sessions per week
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — 12 weeks : 5 sessions per week (1 supervised session at home every month)
  92 weeks : spontaneous training (supervised by phone every month)

SUMMARY:
The study was designed to test the following hypotheses:

Main Objective:

To compare the level of spontaneous physical activity at 3 months after re-entrainment by multi-site electrical stimulation (m-ES), measured by actigraphy over 7 days, compared to conventional care (lifestyle and dietary advice and placebo (simulated) electrostimulation) (control arm).

Secondary Objectives:

To compare the metabolic, inflammatory, cardiovascular and functional parameters, physical activity, quality of life and quality of sleep, at 3 months and at 2 years in the two groups.

Design:

We will conduct a multicenter controlled study vs. reference care with randomization into two parallel groups and double-blind (placebo electrostimulation). Patients will have the ES material available at home and will be supervised by monthly visits over 3 months and by telephone follow-up for two years. The study size calculation is based on physical activity, the percentage of lean body mass and arterial stiffness measured in the OBEX study (NCT01155271).

This project will determine whether the training strategy is effective for increasing physical activity and/or in inducing significant metabolic and cardiovascular effects in these patients after 2 years. In addition, it provides a solid base of investigation for the study of the interactions between muscle contraction and cardio-metabolic health with greater precision.

DETAILED DESCRIPTION:
Obesity and sleep apnea syndrome lead to metabolic troubles and increasing cardiovascular risk. Furthermore, both diseases are associated with reduced exercise tolerance.

For many patients with morbid obesity, the implementation of physical activity programs remains difficult for several reasons including the level of disability and psychosocial causes (the scrutiny of others, depression and poorly adapted equipment).

Main hypothesis: Neuromuscular electrostimulation is a way to increase spontaneous physical activity (PA) in treated apneic obese patients with low spontaneous physical activity

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with BMI > 35 kg/m²
* Continuous Positive Airway Pressure (CPAP) treatment and > 4h observance per night to the patient with OSAS (obstructive sleep apnoea syndrome)
* Patients who give written consent
* Patients who subscribed social insurance

Exclusion Criteria:

* Cardiovascular or respiratory failure discovered at the moment of the inclusion in the study
* Contraindication to exercise
* Pregnant or breast-feed woman
* Patients under guardianship
* Imprisoned patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | After a period of monthly supervised training program by neuromuscular electrical stimulation at home (12th wk)
  * Number of steps per day
  * Number of MET (metabolic equivalent of task) per day

SECONDARY OUTCOMES:
Changes in body composition | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and during a period of spontaneous training (48 th, 72 th, 96 th week)
  Fat mass and fat-mass index as assessed by impedancemetry measurements
Change in arterial stiffness | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and during a period of spontaneous training (48 th, 72 th, 96 th week)
  Pulse wave velocity
Change in endothelial function | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and after a period of spontaneous training (92th week )
  Peripheral arterial tone (RH-PAT)
Change in plasmatic biomarkers | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and after a period of spontaneous training (92th week )
  Oxidative stress and inflammatory blood parameters
Change in quality of life | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and after a period of spontaneous training (92th week )
  SF-12 questionnaire
Number of cardiovascular events per year | Every year from the 1st to the 2th year
  Questionnaire sent to the patient by mail
Change in other parameters of physical activity | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and during a period of spontaneous training (48 th, 72 th, 96 th week)
  Energy expenditure (total and during daily activities)
Change in sleep quality | After a period of monthly supervised training by neuromuscular electrical stimulation at home (12th wk) and during a period of spontaneous training (48 th, 72 th, 96 th week)
  Lying and sleep duration

CONTACTS AND LOCATIONS:
Overall Officials: Renaud TAMISIER, Pr, Principal Investigator — Laboratoire EFCR, CHU de Grenoble, 38043, Grenoble, France
Locations (3):
- France (3):
  - Hôpital Universitaire de Grenoble, Grenoble
  - Hôpital universitaire de Lyon, Lyon
  - Hôpital universitaire de Saint Etienne, Saint-Etienne